CLINICAL TRIAL: NCT01370239
Title: A Multicenter Phase II Study of Treatment With Hu3S193 in Women With Advanced Breast Cancer That Progressed After Hormonal Therapy
Brief Title: HumanaH - Hu3s193 in the Treatment of Advanced Breast Cancer After Hormonal Therapy
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: futility
Sponsor: Instituto do Cancer do Estado de São Paulo (Other)
Collaborators: Fundação Faculdade de Medicina (Other); Recepta Biopharma (Industry)
Responsible Party: Principal Investigator, Paulo Marcelo Gehn Hoff, FACP MD PhD, Full Professor, Instituto do Cancer do Estado de São Paulo
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 52/2009
Record Dates: First submitted 2011-05-25; First posted 2011-06-09 (Estimated); Last update posted 2019-10-11 (Actual); Status verified 2019-10

CONDITIONS: Breast Cancer
Keywords: monoclonal antibody; Lewis; breast cancer
MeSH Terms: conditions — Breast Neoplasms | interventions — Hu3S193 monoclonal antibody

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Hu3S193 (Experimental): Single arm
  Interventions: Biological: Hu3S193

INTERVENTIONS:
Biological: Hu3S193 — Patients will receive weekly intravenous doses of 20 mg/m2 of the antibody Hu3S193. The infusion will take 60 ± 10 minutes. The antibody should be diluted in 500 mL of normal saline.

SUMMARY:
The humanized monoclonal antibody against Lewis Y antigen (Hu3S193) has been demonstrated to be safe in previous studies and has also been indicated as potential intervention in breast cancer. The study of this new agent in advanced breast cancer may contribute to the development of new strategies for patients that progressed after hormonal treatment.

DETAILED DESCRIPTION:
This is a national study, open label, single arm, phase II study which will be conducted in seven centers in Brazil. The study will be coordinated by the INSTITUTO DO CÂNCER DO ESTADO DE SÃO PAULO in collaboration with RECEPTA Biopharma. The study is funded by the CONSELHO NACIONAL DE DESENVOLVIMENTO CIENTÍFICO E TECNOLÓGICO (CNPq). Before any procedure relating to the study, patients must read and sign the informed consent (IC). The inclusion of patients begin immediately after regulatory approval and is expected to end after reaching the number of patients. The follow-up term will last at least 24 months for each patient included, unless limited by death, loss to follow up or withdrawal of informed consent. A total of 60 patients will be recruited in this study. The eligible patients must be 18 or older, confirmed diagnosis of breast cancer with locally advanced or metastatic progression after one or two lines of previous hormone treatment, confirmation of Lewis antigen expression -as assessed by central laboratory, measurable or evaluable disease and adequate organ function. Patients will receive weekly intravenous doses of the antibody Hu3S193 until disease progression, unacceptable toxicity, withdrawal of consent or the investigator's decision, whichever occurs first. The study's primary endpoint is the clinical benefit rate.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of breast cancer with locally advanced or metastatic (stages IIIB, IIIC or IV according to TNM classification), confirmed histologically with no intention to curative treatment by radiotherapy or surgery;
* Clinical or radiological progression after one or two lines of previous hormone treatment, including adjuvant treatment;
* Positive for ER and / or PR expression documented by IHC;
* Confirmed expression of Lewis Y antigen by IHC;
* Presenting the performance status of 0 or 1 according to Eastern Cooperative Oncology Group (ECOG);
* Have a measurable or evaluable disease by Response of Evaluation Criteria in Solid Tumors (RECIST);
* Adequate organ function, assessed by laboratory tests obtained at least 2 weeks before the first day of treatment and within the following parameters:

absolute neutrophil count ≥ 1.5 x 109 / L; platelet count ≥ 100 x 109 / L; serum bilirubin ≤ 2.0 mg / dL; AST/ALT ≤ 2.5 x upper limit of normal; serum creatinine ≤ 2.0 mg / dL;

* Expected survival > 12 weeks;
* In patients with childbearing potential: Negative pregnancy confirmed by test done 21 days before the date of study treatment initiation;
* Willingness and ability to comply with the protocol for the duration of the study.

Exclusion Criteria:

* Patients subjected previously to more than two lines of hormonal therapy, including adjuvant treatment;
* Presenting the amplification or overexpression of HER-2;
* Systemic corticosteroids or immunosuppressive agents used concomitantly with the study or have used systemic corticosteroids or immunosuppressants in the last 14 days before the first dose of the investigational drug;
* Visceral metastatic disease with life-threatening (as defined by extensive liver involvement), or symptomatic pulmonary lymphangitic carcinomatosis or any degree of cerebral or leptomeningeal involvement;
* Previous or current history of clinically significant cardiac disease (class III or IV according to New York Heart Association);
* Clinically significant arrhythmia;
* History of myocardial infarction within the last 6 months;
* Previous or current history of other severe diseases (eg, severe ascites requiring repeated drainage, active infections requiring antibiotics, bleeding, inflammatory bowel disease or chronic diseases that may interfere with obtaining accurate results of the study);
* Previous chemotherapy for metastatic disease (adjuvant chemotherapy is acceptable, if more than four weeks between its completion and inclusion in the study;
* Radiotherapy within 4 weeks before inclusion in the study or with no recovery from the toxic effects of radiotherapy when done up to 6 weeks before inclusion in the study, except for palliative radiotherapy for bone metastases involving <25 % bone marrow;
* Treatment with biological agents, immunotherapy or surgery within 4 weeks before inclusion in the study or with no recovery from the toxic effects of these treatments when made until six weeks prior to study entry (prior treatment with bisphosphonates is allowed, it can be continued after inclusion in the study);
* Any investigational agent treatment within 12 months prior to study entry, unless the investigator considers that the participation in the study may benefit the patient;
* Previous or current history of another type of tumor, excluding skin cancer, melanoma, in situ cervix carcinoma or in situ ductal carcinoma or lobular breast if properly treated;
* Uncontrolled hypercalcemia (defined as total calcium> 11.5 mg / dL)

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 23 (Actual)
Dates: Start 2013-11; Primary Completion 2015-10 (Actual); Study Completion 2018-05-25 (Actual)

PRIMARY OUTCOMES:
Complete response, partial response or stable disease. | more than 24 weeks
  The primary efficacy analysis will be done through the clinical benefit rate, as defined by the proportion of patients achieving best response, complete response, partial response or stable disease for more than 24 weeks

SECONDARY OUTCOMES:
Response rate | 24 weeks after patient discontinuation (at minimum)
  from inclusion until disease progression or death
Non progression rate | 24 weeks after patient discontinuation (at minimum)
  From patient inclusion until disease progression or death - evaluated radiologically by CT
Overall survival | 24 weeks after patient discontinuation (at minimum) or until death
  until death
Progression free survival | until disease progression or 24 weeks after patient discontinuation (at minimum)
  Evaluated radiologically by CT
Assessment of any sign, symptom or undesirable medical condition that occurs after the first administration of the investigational agent | Until disease progression or 30 days after patient discontinuation

CONTACTS AND LOCATIONS:
Overall Officials: PAULO MG HOFF, MD Professor, Study Director — INSTITUTO DO CÂNCER DO ESTADO DE SÃO PAULO; SERGIO V SERRANO, MD, Study Director — HOSPITAL DO CÂNCER DE BARRETOS
Locations (7):
- Brazil (7):
  - Universidade Federal Do Ceará, Fortaleza, Ceará
  - PONTIFíCIA UNIVERSIDADE CATÓLICA DO RIO GRANDE DO SUL, Porto Alegre, Rio Grande do Sul
  - Hospital Do Câncer de Barretos, Barretos, São Paulo
  - Universidade Federal de Goias, Goiás
  - Instituto Nacional Do Câncer, Rio de Janeiro
  - Instituto Do Câncer Do Estado de São Paulo, São Paulo
  - Hospital Sirio Libanes, São Paulo

REFERENCES:
- [Derived] Testa L, Mano M, Arai RJ, Bonadio RC, Serrano SV, Zorzetto MMC, Crocamo S, Smaletz O, Freitas-Junior R, Hoff PM. Phase II trial of humanized anti-Lewis Y monoclonal antibody for advanced hormone receptor-positive breast cancer that progressed following endocrine therapy. Clinics (Sao Paulo). 2021 Oct 11;76:e3146. doi: 10.6061/clinics/2021/e3146. eCollection 2021. PMID 34644735
- See also: COORDINATING CENTER — http://www.icesp.org.br/
- See also: FUNDED BY CONSELHO NACIONAL DE DESENVOLVIMENTO CIENTÍFICO E TECNOLÓGICO — http://www.cnpq.br/